CLINICAL TRIAL: NCT02166112
Title: The Permacol Dutch Cohort Study
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Amphia, Breda, the Netherlands (Unknown); Catharina Ziekenhuis Eindhoven (Other); Franciscus, Roosendaal, the Netherlands (Unknown); Groene Hart, Gouda, the Netherlands (Unknown); Havenziekenhuis (Other); Lievensberg, Bergen op Zoom, the Netherlands (Unknown); Medical Center Haaglanden (Other); MC Leeuwarden, Leeuwarden, the Netherlands (Unknown); Meander MC, Amersfoort, the Netherlands (Unknown); Maastricht University Medical Center (Other); Nij Smellinghe, Drachten, the Netherlands (Unknown); OLVG, Amsterdam, the Netherlands (Unknown); Orbis MC, Sittard, the Netherlands (Unknown); Reinier de Graaf Groep (Other); Rijnstate, Arnhem, the Netherlands (Unknown); Spaarne ziekenhuis, Hoofddorp, the Netherlands (Unknown); Tergooi ziekenhuizen, Hilversum, the Netherlands (Unknown); The Elisabeth-TweeSteden Hospital (Other); UMC Groningen, Groningen, the Netherlands (Unknown); UMC Utrecht, Utrecht, the Netherlands (Unknown); VieCuri, Venlo, the Netherlands (Unknown); Waterland, Purmerend, the Netherlands (Unknown); Zuyderland Medisch Centrum, Sittard-Geleen, the Netherlands (Unknown)
Responsible Party: Principal Investigator, Ruth Kaufmann, MD, PhD fellow, Erasmus Medical Center
Other Study IDs: Permacol Dutch Cohort Study
Record Dates: First submitted 2014-06-10; First posted 2014-06-18 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Hernia of Abdominal Wall; Biologic Implant; Infected Hernioplasty Mesh
Keywords: Hernia of Abdominal Wall; Biologic implant; Infected Hernioplasty Mesh
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Permacol mesh placement: No intervention performed
  Interventions: Procedure: Permacol mesh placement

INTERVENTIONS:
Procedure: Permacol mesh placement — All patients were treated for a complex abdominal wall hernia by implantation of Permacol mesh. This intervention took place before patients were included in the cohort.

SUMMARY:
Incisional hernia is the most frequently seen long term complication in surgery causing much morbidity and even mortality in patients. Despite studies on the optimal closing technique for laparotomies, the risk for incisional hernia after midline incision remains about 5-20 %. It has been established that implementing a mesh reduces recurrence of the incisional hernia but still the results of repair are often disappointing. Incisional hernias can become increasingly complex due to complicated abdominal wall defects caused by a disturbed anatomy, fistulas, burst abdomen, wound and mesh infections. In these cases it is not save to repair the incisional hernia by means of a synthetic mesh and other augmentation tools need to be implemented.

In the recent years the use of biological meshes has been gaining popularity. Recent reports of the use of collagen-based prosthesis have suggested that they support new vessel growth, do not excite a significant foreign body reaction, form fewer adhesions, are well incorporated into host tissues with minimal wound contraction, and can be used in grossly contaminated wounds with fewer infective complications. Biologic meshes are harvested from a source tissue and processed for medical use but they vary widely in their processing methods. They include tissues of human or animal origins, both chemically cross-linked and non cross-linked processes, and submucosal, pericardial, or dermal tissue sources. Current studies investigating the effectiveness of these meshes are small and have short periods of follow-up. These shortcomings can be explained to high cost of the meshes and unclear indication when to use a biological mesh.

The aim of this study is investigate the short and long term effects of the Permacol© biological mesh. Also the investigators will be inquiring why a biologic mesh was used, what is the true indication to use a biological mesh.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Complicated abdominal wall hernia repair
* Permacol© mesh implantation

Exclusion Criteria:

* No signed informed consent
* Operation other than Complicated abdominal wall hernia repair
* Implant other than Permacol© mesh implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The design of the trial will be a cross sectional cohort study. We will be gathering information from all the centers in the Netherlands who have used the Permacol© mesh in the past to treat complicated abdominal wall defects. Patients will be asked to return to the hospitals outpatient clinic. A total of around 70 patients will be included into the study.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Incisional Hernia recurrence | One and two year after initial operation
  This parameter will be assessed by taking a history of the patient and assessing operation room reports.

SECONDARY OUTCOMES:
Mesh explantations | Anytime after abdominal wall reconstruction with Permacol until two years after operation
  This parameter will be assessed by taking a history of the patient and assessing operation room reports.
Postoperative complications | All postoperative complications are assessed until two years after initial operation
  This parameter will be assessed by taking a history of the patient and assessing patient reports and operation room reports.
Additional "abdominal wall repair" operations | After initial abdominal wall reconstruction with Permacol until two years after initial operation
  This parameter will be assessed by taking a history of the patient and assessing patient reports and operation room reports.
Indication of Permacol usage | Perioperatively
  The indication for usage of Permacol was noted just before or just after operation.
Quality of Life | A year or longer after initial abdominal wall reconstruction until two years after initial operation
  This parameter will be assessed various questionnaires (ShortForm-36, EuroQOL (EQ-5D-5L), and Body Image Questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Kaufmann, MD, Study Chair — Erasmus Medical Center
Locations (24):
- Netherlands (24):
  - Meander MC, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Rijnstate, Arnhem
  - Lievensberg, Bergen op Zoom
  - Amphia, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Nij Smellinghe, Drachten
  - Catharina, Eindhoven
  - Groene Hart, Gouda
  - UMC Groningen, Groningen
  - Atrium MC, Heerlen
  - Tergooi ziekenhuizen, Hilversum
  - Spaarne ziekenhuis, Hoofddorp
  - MC Leeuwarden, Leeuwarden
  - MUMC+, Maastricht
  - Waterland, Purmerend
  - Franciscus, Roosendaal
  - Erasmus University Medical Center, Rotterdam
  - Havenziekenhuis, Rotterdam
  - Orbis MC, Sittard
  - MC Haaglanden, The Hague
  - TweeSteden, Tilburg
  - UMC Utrecht, Utrecht
  - VieCuri, Venlo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaufmann R, Timmermans L, van Loon YT, Vroemen JPAM, Jeekel J, Lange JF. Repair of complex abdominal wall hernias with a cross-linked porcine acellular matrix: cross-sectional results of a Dutch cohort study. Int J Surg. 2019 May;65:120-127. doi: 10.1016/j.ijsu.2019.03.023. Epub 2019 Apr 1. PMID 30946996